CLINICAL TRIAL: NCT03838107
Title: Identifying Markers of Trajectory in Pediatric Complex Regional Pain Syndrome
Brief Title: Markers of Trajectory in Pediatric CRPS
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-1565
Record Dates: First submitted 2018-08-24; First posted 2019-02-12 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Complex Regional Pain Syndromes
Keywords: pediatric complex regional pain syndrome; fMRI; psychosocial; quantitative sensory testing; markers
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Inpatients: Observation and measure of trajectory of recovery in CRPS. This group will include children diagnosed with CRPS and undergoing regular therapy at the inpatient FIRST clinic at CCHMC and one of their parents or legal guardian.
  Interventions: Behavioral: observation and measure of trajectory of recovery in CRPS
- Outpatients: Observation and measure of trajectory of recovery in CRPS. This group will include children diagnosed with CRPS and undergoing regular therapy at the outpatient Pain Management Center at CCHMC and one of their parents or legal guardian.
  Interventions: Behavioral: observation and measure of trajectory of recovery in CRPS
- Healthy Controls: For comparison purposes, healthy controls and one of their parents or legal guardian will be enrolled in this study as well.
  Interventions: Behavioral: observation and measure of trajectory of recovery in CRPS

INTERVENTIONS:
Behavioral: observation and measure of trajectory of recovery in CRPS — Child participants enrolled in this study will undergo three sessions, which will include psychosocial measures, brain imaging, and quantitative sensory testing. Parent participants will also complete three sessions, which only include psychosocial measures.

SUMMARY:
Complex Regional Pain Syndrome (CRPS) is a severe and complex chronic pain condition in children. Many psychosocial factors impact its development and recovery. CRPS has a strong central component, which is reflected by structural and functional changes in the brain. However, the interaction between these cerebral changes and trajectory of recovery has been seldom investigated to date. Furthermore, interactions between cerebral changes and psychosocial factors, which might affect trajectory of recovery, are unknown. The aim of this study is to identify the psychosocial factors and cerebral changes that predict the trajectory of recovery from CRPS.

Children between the ages of 10 and 17 years will be enrolled with one of their parents or legal guardians for this study. Three populations will be recruited: patients with CRPS undergoing treatment at the Functional Independence Restoration Program (FIRST), patients with CRPS undergoing treatment at the Pain Management Center and matching healthy controls. Participants will undergo three sessions: the first session will be scheduled immediately before or as soon as possible at the beginning of the patients' treatment; the second session will take place at the end of the patients' treatment; the last session will be scheduled six months post-treatment. The timing of the sessions of the healthy participants will follow a schedule similar to the FIRST patients. Each session will last approximately three hours and include acquisition of psychosocial, psychophysical, and brain imaging data in the child participants, as well as acquisition of psychosocial data in the parent participants.

DETAILED DESCRIPTION:
This is a basic science investigation of potential psychosocial, sensory, and brain markers predicting trajectory of short-term and long-term recovery in pediatric CRPS following both inpatient and outpatient treatment.

The usual inpatient treatment lasts on average three weeks and includes physical, occupational, and recreational therapy, as well as psychotherapy, while patients keep their regular pharmacological treatment. The usual outpatient treatment lasts on average several months and includes physical therapy and psychotherapy, in addition to pharmacotherapy. For both inpatients and outpatients, the primary anti-neuropathic pharmacotherapy typically includes gabapentin, pregabalin, or amitriptyline, or, less frequently, duloxetine. It is important to note that this study is not designed to investigate the efficacy of treatment per se, instead it aims to predict trajectory during the course of treatment as usual. This study is primarily mechanistic and does not include any intervention or modification of treatments. Therefore, patients, who are scheduled for regular inpatient or outpatient treatment of CRPS, are free to refuse to enroll without any consequences for the scheduled treatment.

The investigated markers will be assessed in patients undergoing inpatient or outpatient treatments. To define potentially relevant markers, measurements in patients will be compared to the same measurements in healthy children. For this purpose, participants will undergo a testing session just before the beginning of their treatment or as close as possible from the beginning of their treatment.

To establish the influence of potential markers on short-term recovery, patients will undergo an additional session upon completion of their treatment. To investigate the effect of the previously defined markers on long-term recovery, patients will complete a third session at six months after treatment. For comparison purposes, healthy control children will undergo sessions following the same schedule as the patients. To assess the association between symptoms of CRPS in children and social environment, at least one parent of each enrolled child will be asked to complete three sessions following the same schedule as their child.

Each testing session will include self-reported questionnaires for the children and their parents and a brain imaging session for the children.

ELIGIBILITY:
Inclusion Criteria:

All Children:

* Age between 10 and 17 years old
* Fluent in English

Inpatients:

* Diagnosis of CRPS
* Former unsuccessful treatment for CRPS
* Scheduled for or beginning the usual inpatient treatment for CRPS at the FIRST clinic at CCHMC.

Outpatients:

* Diagnosis of CRPS
* Scheduled for or beginning the usual outpatient treatment for CRPS at the pain management clinic

Healthy children:

- No diagnosis of chronic pain.

Parents:

* Fluent in English
* Child participating in the study

Exclusion Criteria:

All child participants:

* Weight/size incompatible with MRI scanner
* Identification of brain, neurologic, or severe psychiatric abnormalities beyond those normally associated with chronic pain.
* Documented developmental delays or impairment
* Any MRI contra-indication, including
* Braces, stents, clips, pace-maker or other metal implants affecting the safety of the participants in the scanner and/or the quality of the images
* pregnancy
* claustrophobia

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants to this study may be part of one of the following groups: children diagnosed with CRPS undergoing inpatient treatment at the FIRST clinic (CCHMC), children diagnosed with CRPS underdoing outpatient treatment at the pain management clinic (CCHMC or comparable outpatient programs), or healthy children. The investigator's groups will be matched as well as possible for BMI, sex, and age. In addition, one parent will be recruited with each child.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2018-08-27 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
changes in pain perception | before treatment, at the end of the treatment (an average of 4 weeks for inpatients and 3 months for outpatients after session 1), and 6-month post treatment for patients; 1 month after session 1 and 6 months after session 2 for healthy participants
  changes in ratings of spontaneous pain intensity and unpleasantness assessed on non-numerical visual analog scales, ranging from 'no pain sensation'/'not at all unpleasant' to 'most intense pain sensation imaginable'/'most unpleasant imaginable'
Changes in functional disability | before treatment, at the end of the treatment (an average of 4 weeks for inpatients and 3 months for outpatients after session 1), and 6-month post treatment for patients; 1 month after session 1 and 6 months after session 2 for healthy participants
  Changes in scores on the self-reported Functional Disability Inventory investigates disabilities associated with pain which might impact on everyday functioning of children. It includes 15 questions assessing the children's capacity to perform everyday tasks, such as doing chores, walking, or eating regular meals. Participants evaluate their capacity to perform these tasks on Likert-type scale, ranging from "No Trouble" to "Impossible".

SECONDARY OUTCOMES:
Changes in functional Magnetic Resonance Imaging (fMRI) BOLD (Blood Oxygenation Level Dependent) and pCASL (pseudo-Continuous Arterio-Spin Labeling) resting-state and task-related brain signal | before treatment, at the end of the treatment (an average of 4 weeks for inpatients and 3 months for outpatients after session 1), and 6-month post treatment for patients; 1 month after session 1 and 6 months after session 2 for healthy participants
  fMRI BOLD and PCASL will be used to measure changes in brain activation at rest and during a multisensory task
changes in fMRI BOLD and pCASL resting-state functional connectivity | before treatment, at the end of the treatment (an average of 4 weeks for inpatients and 3 months for outpatients after session 1), and 6-month post treatment for patients; 1 month after session 1 and 6 months after session 2 for healthy participants
  fMRI BOLD and pCASL will be used measure of changes in functional connectivity at rest
changes in DTI (Diffusion Tensor Imaging) structural connectivity | before treatment, at the end of the treatment (an average of 4 weeks for inpatients and 3 months for outpatients after session 1), and 6-month post treatment for patients; 1 month after session 1 and 6 months after session 2 for healthy participants
  Diffusion tensor imaging will be used to measure changes in structural connectivity

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Coghill, PhD, Principal Investigator — Children's Hospital, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-12): https://cdn.clinicaltrials.gov/large-docs/07/NCT03838107/Prot_SAP_000.pdf